CLINICAL TRIAL: NCT04992312
Title: An Open-Label, Multi-Center, Single-Dose Study to Assess the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of Nasal Glucagon in Pediatric Patients With Type 1 Diabetes Aged 1 to <4 Years
Brief Title: A Study of Nasal Glucagon (LY900018) in Pediatric Participants With Type 1 Diabetes
Acronym: RescuiNGkids
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17449; I8R-MC-IGBO (Other: Eli Lilly and Company); 2021-006088-61 (EudraCT Number)
Record Dates: First submitted 2021-08-04; First posted 2021-08-05 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Type 1 Diabetes
Keywords: Severe Hypoglycemia; Nasal Powder; Hypoglycemia Rescue Therapy; Ready to use Glucagon
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 3 milligram (mg) Nasal Glucagon (Experimental): Participants received a single dose of 3 mg glucagon powder administered intranasally on day 1.
  Interventions: Drug: Glucagon Nasal Powder [Baqsimi]

INTERVENTIONS:
Drug: Glucagon Nasal Powder [Baqsimi] — Administered intranasally
  Other Names: LY900018; Baqsimi

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of a study drug called nasal glucagon (Baqsimi) in pediatric participants with type 1 diabetes (T1D) aged 1 to less than 4 years. Blood tests will be performed to check how much nasal glucagon gets into the bloodstream. Blood sugar will also be measured to understand the effect of the drug on blood sugar levels. The study consists of a screening period up to 35 days before dosing, 1 day when a dose of nasal glucagon will be given and then 2 telephone follow up calls; first follow-up call on the day after the nasal glucagon was given and second call about one week after nasal glucagon was given. The study will last up to 9 days, not including the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Have a Type 1 Diabetes diagnosis for at least 6 months
* Have been receiving insulin therapy via multiple daily injections or using an insulin pump and have been stable for at least 3 months prior to screening
* Have a HbA1c level of ≤ 9.5% at screening
* Have sufficient venous access for collection of blood samples
* Have good general health, apart from their Type 1 diabetes, with no prior history of choanal atresia, nasal/pharyngeal blockage or nasal anomaly

Exclusion Criteria:

* Have a presence or history of glucagon hypersensitivity
* Have a history of pheochromocytoma
* Have a history of epilepsy or seizure disorder
* Have 1 or more congenital anomalies to the anatomy of the nose, or require changes to the anatomy of the nose
* Are using closed-loop insulin therapy, unless such a device is set to 'open loop/manual' mode on the day of the dosing visit
* Have an episode of severe hypoglycemia or have had glucagon administered , during the 3 months prior to the screening visit and no severe hypoglycemia between the screening and dosing visit

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-11-05 (Actual); Study Completion 2023-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- United States (8):
  - Nemours Childrens Clinic, Jacksonville, Florida
  - St. Luke's Regional Medical Center, Boise, Idaho
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - UBMD Pediatrics, Buffalo, New York
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of Nasal Glucagon (LY900018) in Pediatric Participants With Type 1 Diabetes (RescuiNGkids) — https://trials.lillytrialguide.com/en-US/trial/3M5oZzkbDqRlSiqf7KNpeL

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3 Milligram (mg) Nasal Glucagon
Started | 7
Received at Least One Dose of Study Drug | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- 3 mg Nasal Glucagon: Participants received a single dose of 3 mg glucagon powder administered intranasally on day 1.
Arm/Group | 3 mg Nasal Glucagon
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.98 (0.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Treatment-Emergent Adverse Event(s) (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A TEAE is defined as an adverse event which occurs post-dose or which is present prior to dosing and becomes more severe post-dose. An SAE is any AE from the study that results in 1 of the following: Death, initial or prolonged inpatient hospitalization, a life-threatening experience (i.e., immediate risk of dying), persistent or significant disability/incapacity, congenital anomaly/birth defect, important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent 1 of the other outcomes listed in the definition above. The number of participants with one or more TEAEs, SAEs considered by the investigator to be related to study drug administration is reported here. A summary of SAEs and other non-serious AEs, regardless of causality is located in the Reported Adverse Events section of this record.
Time Frame: Baseline to Day 9
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg Nasal Glucagon
Number analyzed (Participants) | 7
Participants
  TEAEs | 5
  SAEs | 0

2. Secondary Outcome: Pharmacodynamics (PD): Change From Baseline in Maximum Observed Blood Glucose (BGmax)
Description: Change from baseline in BGmax was measured to investigate the PD effect of nasal glucagon on blood glucose level following 3 mg nasal glucagon administration on day 1. Baseline is defined as Day 1 pre-dose. The BGmax on Day 1 was determined using plasma samples collected pre-dose, 10, 30, 60, and 90 minutes post nasal glucagon dose.
Time Frame: Baseline, Day 1 (pre-dose, 10, 30, 60, 90 minutes post-dose)
Population: All participants who received at least one dose of study drug and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | 3 mg Nasal Glucagon
Number analyzed (Participants) | 7
milligrams per deciliter (mg/dL) | 132.4 (52.4)

3. Secondary Outcome: PD: Absolute BGmax of Nasal Glucagon
Description: PD: Absolute BGmax of Nasal Glucagon
Time Frame: Day 1 (pre-dose, 10, 30, 60, 90 minutes post-dose)
Population: All participants who received at least one dose of study drug and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 3 mg Nasal Glucagon
Number analyzed (Participants) | 7
mg/dL | 242.1 (46)

4. Secondary Outcome: PD: Time of Maximum Observed Blood Glucose (TBGmax) of Nasal Glucagon
Description: PD: TBGmax of Nasal Glucagon
Time Frame: Day 1 (pre-dose, 10, 30, 60, 90 minutes post-dose)
Population: All participants who received at least one dose of study drug and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 3 mg Nasal Glucagon
Number analyzed (Participants) | 7
minutes | 55.6 (20.9)

5. Secondary Outcome: PD: Area Under the Concentration Versus Time Curve (AUC) of Blood Glucose
Description: AUC from time 0 to the last measured concentration of blood glucose at 90 minutes [AUC(0-90)] is reported.
Time Frame: Day 1 (pre-dose, 10, 30, 60, 90 minutes post-dose)
Population: All participants who received at least one dose of study drug and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: milligram*minute per deciliter (mg*m/dL)
Arm/Group | 3 mg Nasal Glucagon
Number analyzed (Participants) | 7
milligram*minute per deciliter (mg*m/dL) | 18200 (3000)

6. Secondary Outcome: Pharmacokinetics (PK): AUC of Nasal Glucagon
Description: PK: AUC of Nasal Glucagon
Time Frame: Day 1 (10, 30, 60 minutes post-dose)
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram*hour per milliliter (pg*hr/mL)
Arm/Group | 3 mg Nasal Glucagon
Number analyzed (Participants) | 7
picogram*hour per milliliter (pg*hr/mL) | 1560 (25.3)

ADVERSE EVENTS:
Time Frame: Baseline to Day 9
Description: All participants who received at least one dose of study drug.
Arm/Group | 3 mg Nasal Glucagon
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 5/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mg Nasal Glucagon (N=7)
Eye pruritus (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Post-tussive vomiting (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT04992312/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT04992312/SAP_001.pdf